CLINICAL TRIAL: NCT04667832
Title: Ankle-brachial Index a Simple and Inexpensive Screening Test for Coronary Artery Disease (ABI Goes Beyond the Foot)
Brief Title: ABI for Screening of Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Kojuri, Professor, Shiraz University of Medical Sciences
Other Study IDs: IR.SUMS.MED.REC.1398.437
Record Dates: First submitted 2020-12-04; First posted 2020-12-16 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; vitamin D deficiency
MeSH Terms: conditions — Coronary Artery Disease; Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- abnormal ABI: those patients with ankle brachial index ( ABI) less than 0.9
  Interventions: Diagnostic Test: selective coronary artery angiography
- normal ABI: Those patients with ankle brachial index more than 0.9
  Interventions: Diagnostic Test: selective coronary artery angiography

INTERVENTIONS:
Diagnostic Test: selective coronary artery angiography — Radial approach, invasive selective coronary angiography with selective contrast injection and filming in coronary arteries

SUMMARY:
Large population cross sectional study between 2019-2020 for 4207 new patients that refer to professor Kojuri cardiovascular clinic in shiraz, Iran, was conducted. Patients were undergone selective coronary angiography from radial artery approach by an expert interventional cardiologist. ABI were measured for all patients. ABI ratio was compared with the results of coronary angiography for patients who underwent coronary angiography to measure specificity and sensitivity.

DETAILED DESCRIPTION:
This cross-sectional study was conducted between 2019 -2020. Inclusion criteria was all of the new patients who referred to Professor Kojuri cardiovascular clinic in Shiraz, Iran (Iran, Fars Province, Shiraz, Niayesh Boulevard kojurij@yahoo.com, http://kojuriclinic.com ) Exclusion criteria was Patients with DVT, Lower extremity wound that cause severe pain and patients who were unable to remain supine. Patients with ABI more than 1.4 were also Excluded.

Complete history and physical exam were taken from the patients and risk factors such as smoking, hypertension, dyslipidemia, diabetes mellitus, age and gender were considered. We checked triglyceride, total cholesterol, LDL cholesterol, HDL cholesterol, HbA1c and High sensitive CRP (Hs-CRP) for all patients. Blood pressure was measured and electrocardiography (EKG) was taken for all patients.

Dyslipidemia were defined as high total or LDL cholesterol, high triglyceride or low HDL cholesterol. Diabetes diagnosis were based on 2019 American diabetes association guideline. Hypertension were defined according to American heart association 2017.

Triglyceride more than 200, Total Cholesterol more than 200, LDL more than 100, HDL less than 40 for men and less than 50 for women, HbA1c more than 6.5 and Hs-CRP more than 2 were considered abnormal. Patients with Hs-CRP more than 10 were excluded due to possibility of Acute inflammation. Smoking were defined as regular tobacco smoking or past history of smoking within 3 months before their visit.

No evidence of abnormal findings in non-invasive studies were considered absence of CAD. Patients with strongly positive results of noninvasive studies, were undergone selective coronary angiography from radial artery approach by an expert interventional cardiologist. Angiography videos were reviewed by a team of expert cardiologists. Based on the results of coronary angiography, patients were classified as mild proven CAD with stenosis less than 50% and severe proven CAD with stenosis more than 50% stenosis.

ABI performed for all patients with Huntleigh Dopplex ABIlity Automatic Ankle Brachial Index System. It was made in Cardiff, United kingdom. This device used Doppler ultrasound for measuring ABI. The appropriate cuffs were selected for patients. Patients were supine 30 minutes before starting test. Ankle and brachial cuffs were attached directly to the patient's skin. Both left and Right ABI were measured. ABI under 0.9 were considered as Abnormal ABI. ABI between 0.9 and 1.4 were assumed as Normal ABI. Patients with both right and left ABI between 0.9 and 1.4 were classified as normal ABI patients. Other patients with at least right or left ABI under 0.9 were considered as abnormal ABI patients. Inter-arm systolic pressure difference was also measured for patients. Inter-arm systolic pressure difference over 10mmhg were considered abnormal.

This study was double-blinded. The team of cardiologists who reported the results of coronary angiography were blinded about the results of patient's ABI. The statisticians also didn't have information about the results of ABI and coronary angiography. For blinding, we used alphabet for each group of patients with or without coronary artery disease. We also used alphabet for normal or abnormal ABI.

For statistical analysis IBM SPSS statistics version 25 was used . Independent sample t test and one-way ANOVA were used for parametric variables. We used Mann-whitney u test and Kruskal-Wallis test for nonparametric data. P value 0.05 were assumed significant.

All of the patients were informed about the details of this research and written consent were obtained from them. Patients who disagreed were excluded from this study

ELIGIBILITY:
Inclusion Criteria:

* patients who referred to Professor Kojuri cardiovascular clinic

Exclusion Criteria:

* Patients with DVT
* Lower extremity wound that cause severe pain
* Patients who were unable to remain supine
* Patients with ABI more than 1.4

Ages: 30 Years to 88 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: About 4207 new patients referred to our cardiovascular clinic. 91 patients were excluded based on the Exclusion criteria. ABI was performed for 4116 patients. There were 2179(52.9%) women and 1937(47.1%) men. The mean age of the patients was 63(30-88).
Sampling Method: Non-Probability Sample
Enrollment: 4207 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
coronary artery disease | 1 year
  lesion more than 50% in selective coronary angiography

SECONDARY OUTCOMES:
Hs-CRP | 1 year
  level of serum high sensitivity CRP, which ids abnormal with more than 2 mg/L

CONTACTS AND LOCATIONS:
Locations (1):
- Professor kojuri cardiology clinic, Shiraz, Outside of the US, Iran

IPD SHARING:
Plan to Share IPD: No
not till publication